CLINICAL TRIAL: NCT00174486
Title: A Double Blind, Placebo Controlled, Parallel Group, Multicenter Study To Assess The Duration Of Action, Safety And Toleration Of Differing Doses and Combinations Of Immediate and Modified Release Formulations Of UK-369,003 and Cialis Compared To Placebo In Adult Male Subjects With Erectile Dysfunction
Brief Title: Assessment Of Duration Of Action, Safety & Toleration Of UK369,003 and Cialis In Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3711030
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2005-11

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

INTERVENTIONS:
Drug: UK0369,003
Drug: Cialis (Tadalafil)

SUMMARY:
Assessment of duration of action, safety & toleration of different formulations and doses of UK-369,003 and Cialis in patients with male erectile dysfunction. Patients should have previously been on PDE5 inhibitors and have been respondents to the drug. Duration of treatment is 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Erectile Dysfunction

Exclusion Criteria:

* Alpha blockers and Nitrates of any preparation

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2005-02; Study Completion 2005-06

PRIMARY OUTCOMES:
Assessment of duration of action, safety & toleration of the investigational drug and Cialis

SECONDARY OUTCOMES:
Assess safety & toleration over 4 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer